CLINICAL TRIAL: NCT03570398
Title: A Feasibility Randomised Control Trial to Evaluate the Role of Computed Tomography in Patients With Indeterminate Right Iliac Fossa Pain
Brief Title: Imaging Possible Appendicitis With CT
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016040
Record Dates: First submitted 2018-05-25; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal CT (Other)
  Interventions: Other: unenhanced abdomino-pelvic CT scan
- Abdominal Ultrasound (Other)
  Interventions: Other: abdominal ultrasound

INTERVENTIONS:
Other: unenhanced abdomino-pelvic CT scan — unenhanced abdomino-pelvic CT scan
  Arms: Abdominal CT
Other: abdominal ultrasound — abdominal ultrasound
  Arms: Abdominal Ultrasound

SUMMARY:
Pain in the right lower abdomen is one of the commonest reasons patients present to general surgeons as an emergency. Whether or not such patients have appendicitis is crucial to their assessment. In UK practice, when the diagnosis is unclear, ultrasound scanning (US) is commonly used to investigate the problem. US is very safe but it will only visualise the appendix in the minority of cases. As a result, the sensitivity for diagnosing appendicitis in this setting is probably only 5-30%. Alternatively, computed tomography (CT) is an accurate way of diagnosing appendicitis in over 90% of cases. CT scans are readily available and with modern scanners, high quality images can be achieved with lower radiation doses. Unenhanced scanning avoids the use of contrast media and permits further reductions in ionising radiation exposure.

DETAILED DESCRIPTION:
Pain in the right lower abdomen is one of the commonest reasons patients present to general surgeons as an emergency. Whether or not such patients have appendicitis is crucial to their assessment. In UK practice, when the diagnosis is unclear, ultrasound scanning (US) is commonly used to investigate the problem. US is very safe but it will only visualise the appendix in the minority of cases. As a result, the sensitivity for diagnosing appendicitis in this setting is probably only 5-30%. Alternatively, computed tomography (CT) is an accurate way of diagnosing appendicitis in over 90% of cases. CT scans are readily available and with modern scanners, high quality images can be achieved with lower radiation doses. Unenhanced scanning avoids the use of contrast media and permits further reductions in ionising radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

• Acute presentation with abdominal pain and/or tenderness which is most marked in the right lower abdomen

Exclusion Criteria:

* Age<18
* Age>60
* Pregnancy
* Patients with a firm clinical diagnosis of appendicitis where surgical management is indicated at presentation
* Patients who have undergone CT scanning within the past two months
* Patients with cognitive impairment who would lack capacity to give consent
* Inability to understand written or spoken English
* Patients who have previously undergone appendicectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 years
  As assessed by the rate of refusal to participate amongst eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Peter Davis, MD, Principal Investigator — James Cook University Hospital
Locations (1):
- South Tees Hospitals NHS Foundation Trust, Middlesbrough, United Kingdom